CLINICAL TRIAL: NCT02628769
Title: A Single-center, Double-blind, Randomised, Placebo-controlled Crossover Study to Evaluate the Effect of Solithromycin on Airway Inflammation in Male and Female Patients With Chronic Obstructive Pulmonary Disease
Brief Title: A Study to Evaluate the Anti-inflammatory Effects of Solithromycin in Chronic Obstructive Pulmonary Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Melinta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CE01-204; 2014-003077-42 (EudraCT Number); 14/LO/2066 (Other: NRES Reference Number)
Record Dates: First submitted 2015-12-01; First posted 2015-12-11 (Estimated); Results first posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Solithromycin; Chronic Obstructive Pulmonary Disease; Inflammation; Macrolide
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Inflammation | interventions — solithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Solithromycin (Experimental): 28 day treatment of 400 mg Solithromycin taken once a day.
  Interventions: Drug: Solithromycin
- Placebo (Placebo Comparator): 28 day treatment with placebo taken once per day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Solithromycin
  Other Names: CEM-101
  Arms: Solithromycin
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study examines the potential benefit of a new antibiotic, Solithromycin, for the long-term treatment of Chronic Obstructive Pulmonary Disease (COPD). Solithromycin is hypothesised to work by reducing inflammation in the lungs of patients with COPD. Stable COPD patients will receive treatment with solithromycin for 28 days and comparisons will be made between any effects observed with Solithromycin and a placebo. This will include any changes in inflammatory proteins, lung function and reported symptoms.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a common and debilitating respiratory illness, that kills around 30,000 people annually in the UK. The primary risk factor is cigarette smoking, which causes inflammation in the air passages of the lungs. This inflammation is irreversible and results in progressive lung destruction. Currently, there are no effective anti-inflammatory medications available for COPD.

Inhalers remain the mainstay of regular treatment for COPD. Macrolide antibiotics however, are occasionally used as a supplementary treatment for some patients. They have been shown to be anti-inflammatory. However, concerns exist over the development of bacterial resistance to such antibiotics. Consequently they are not widely prescribed for COPD. Solithromycin is a new macrolide antibiotic, which has been shown to possess superior anti-inflammatory properties. Importantly, bacteria are far less likely to develop resistance to this new medication.

The current study will assess the effect of solithromycin as an anti-inflammatory treatment for COPD. 30 patients will be recruited to receive 28 days of treatment with solithromycin or placebo, followed by a 28 day wash out period (no study medication), before taking a further 28 days of treatment (the medication not taken first time around, i.e. either solithromycin or placebo). This study is a single-centre (Harefield Hospital), double-blind (study team and patient are not told what treatment they are taking), randomised (order in which solithromycin and placebo are taken), placebo-controlled and has a crossover design (subjects take both solithromycin and placebo separately). Sputum, blood and fluid from the nasal lining will be periodically sampled to examine any effect on the levels of inflammatory cells and proteins during the study. Any changes in lung function parameters or symptoms (COPD Assessment Test) will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. History of cigarette smoking >10 pack-years.
2. Post-bronchodilator FEV1/FVC of <0.70 and FEV1 of 30-79% of predicted normal value.
3. Patients on prescribed inhaled corticosteroids can be enrolled.
4. Females of non-childbearing potential: surgically sterile (e.g. tubal ligation) or at least 2 years post-menopausal.
5. Females of childbearing potential (including females less than 2 years post-menopausal) must have a negative pregnancy test at enrollment and must agree to use highly effective methods of birth control (i.e. diaphragm plus spermicide or male condom plus spermicide, oral contraceptive in combination with a second method, contraceptive implant, injectable contraceptive, indwelling intrauterine device, sexual abstinence, or a vasectomized partner) while participating in the study and for 30 days after the last dose of study drug.
6. The patient must be willing and able to comply with all study visits and procedures.
7. The patient must be a suitable candidate for oral therapy and be able to swallow capsules intact.
8. The patient must provide written informed consent.
9. No evidence of active bacterial infection in sputum by qPCR evaluation.

Exclusion Criteria:

1. Acute exacerbation of COPD within the previous 60 days or during the washout period of the study.
2. Any condition that could possibly affect oral drug absorption, e.g. gastroenteritis, status post gastrectomy, status post bariatric surgery.
3. Currently taking medication for HIV, chronic hepatitis B, or hepatitis C virus (HCV) infection.
4. Currently taking theophylline or other xanthine medication.
5. Currently taking warfarin.
6. Known concomitant infection (pulmonary or otherwise) which would require additional systemic antibiotics.
7. QTc greater than 450 msec for males or females as corrected by the Fridericia formula.
8. Current use of drugs known to prolong the QT interval, including Class Ia (quinidine, procainamide) or Class III (amiodarone, sotalol) antiarrhythmics.
9. Concomitant use of drugs, foods, or herbal products known to be moderate to potent inhibitors of CYP3A4 isozymes: oral antifungal agents (e.g. ketoconazole, itraconazole, posaconazole, fluconazole and voriconazole); HIV protease inhibitors (e.g. ritonavir and saquinavir), HCV protease inhibitors (e.g. boceprevir and telaprevir), nefazodone, fluvoxamine, conivaptan, diltiazem, verapamil, aprepitant, ticlopidine, crizotinib, imatinib; grapefruit or grapefruit juice.
10. Any use within the prior 7 days of drugs or herbal products known to be moderate to potent inducers of CYP3A4 isozymes: St. John's Wort, rifampin, rifabutin, anti-convulsants (e.g. phenobarbital, carbamazepine, phenytoin, rufinamide), modafinil, armodafinil, etraverine, efavirenz, bosentan.
11. Required current use of drugs with narrow therapeutic indices that are principally metabolized by CYP3A4 or transported by P-glycoprotein (P-gp), for which a drug interaction with solithromycin could result in higher and possibly unsafe exposures to these drugs: e.g. the P-gp substrates digoxin or colchicine and the CYP3A4 substrates alfentanil, astemizole, cisapride, cyclosporine, dihydroergotamine, ergotamine, fentanyl, midazolam, pimozide, quinidine, sirolimus, tacrolimus, everolimus, and terfenadine).
12. History of organ transplant.
13. Cytotoxic chemotherapy or radiation therapy within the previous 3 months.
14. Known neuromuscular disorder from clinical history (e.g. myasthenia gravis, Parkinson's disease).
15. Known significant renal, hepatic, or hematologic impairment.
16. Women who are pregnant or breast feeding
17. Prior participation in this protocol.
18. Any investigational drugs taken or investigational devices used within 4 weeks before administration of the first dose of the study drug.
19. History of intolerance or hypersensitivity to macrolide antibiotics.
20. Any concomitant condition that, in the opinion of the Investigator, would preclude an evaluation of a response or make it unlikely that the contemplated course of therapy and follow-up could be completed (e.g. life expectancy <30 days).

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-01-05 (Actual); Study Completion 2017-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Barnes, FRS, FMedSci, Principal Investigator — Imperial College London; William Man, MBBS, PhD, Study Chair — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Muscle Lab, Respiratory Medicine, Harefield Hospital, Harefield, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- First Solithromycin, Then Placebo: First 28-day treatment of 400 mg Solithromycin taken once a day, then 28-day treatment with placebo taken once per day.
- First Placebo, Then Solithromycin: First 28-day treatment with placebo taken once per day, then 28-day treatment of 400 mg Solithromycin taken once a day.
Period: First Intervention
Arm/Group | First Solithromycin, Then Placebo | First Placebo, Then Solithromycin
Started | 3 | 3
Completed | 2 | 2
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Period: Wash Out (28 Days)
Arm/Group | First Solithromycin, Then Placebo | First Placebo, Then Solithromycin
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | First Solithromycin, Then Placebo | First Placebo, Then Solithromycin
Started | 2 | 2
Completed | 0 | 1
Not Completed | 2 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participant: All participants cross-over study
Arm/Group | All Participant
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.7 (3)
FEV1 [Mean (Standard Deviation); unit: litre] — Lung function parameter
  litre | 1.29 (0.03)
COPD Assessment Test (CAT) [Mean (Standard Deviation); unit: scores on a scale] — The COPD Assessment Test (CAT) is a questionnaire for people with Chronic Obstructive Pulmonary Disease (COPD). It is designed to measure the impact of COPD on a person's life. The scores from 0-40. Higher scores denote a more severe impact of COPD on a patient's life.
  scores on a scale | 17 (7.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Sputum Neutrophils Per mL at 28 Days
Description: A number of sputum neutrophils per mL after treatment with solithromycin and placebo.
Time Frame: 28 days
Population: Due to the early termination of the study, there were too few subjects and data collected to perform statistical analysis
Measure: Mean (Standard Error); unit: 10^6 cells/ml sputum
Arm/Group | Solithromycin | Placebo
Number analyzed (Participants) | 3 | 4
10^6 cells/ml sputum | 2.47 (0.76) | 5.30 (1.21)

2. Secondary Outcome: Concentrations of Sputum CXCL8 at 28 Days
Description: Concentrations of sputum CXCL8 after treatment with solithromycin and placebo.
Time Frame: 28 days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Solithromycin | Placebo
Number analyzed (Participants) | 3 | 4
ng/ml | 2.99 (0.76) | 4.29 (0.43)

3. Secondary Outcome: Concentrations of Sputum IL-6 Before and After Treatment With Solithromycin and Placebo at 28 Days
Time Frame: 28 days
Population: No data collected for this Outcome due to early termination of the trial
Arm/Group | Solithromycin | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Concentrations of Sputum MPO Before and After Treatment With Solithromycin and Placebo at 28 Days
Time Frame: 28 days
Population: No data collected for this Outcome due to early termination of the trial
Arm/Group | Solithromycin | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Concentrations of Sputum MMP-9 Before and After Treatment With Solithromycin and Placebo at 28 Days
Time Frame: 28 days
Population: No data collected for this Outcome due to early termination of the trial
Arm/Group | Solithromycin | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Concentrations of Sputum MCP-1 Before and After Treatment With Solithromycin and Placebo.
Time Frame: 28 days
Population: No data collected for this Outcome due to early termination of the trial
Arm/Group | Solithromycin | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Concentrations of Sputum TNF-α Before and After Treatment With Solithromycin and Placebo.
Time Frame: 28 days
Population: No data collected for this Outcome due to early termination of the trial
Arm/Group | Solithromycin | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Concentrations of CXCL8 in Nasal Lining Fluid With Solithromycin and Placebo at 28 Days
Time Frame: 28 days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Solithromycin | Placebo
Number analyzed (Participants) | 3 | 4
ng/ml | 1.39 (0.58) | 5.14 (1.6)

9. Secondary Outcome: FEV1 After Treatment With Solithromycin and Placebo at 28 Days
Time Frame: 28 days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: litre
Arm/Group | Solithromycin | Placebo
Number analyzed (Participants) | 3 | 4
litre | 1.13 (0.16) | 1.05 (0.08)

10. Secondary Outcome: R5-R20 After Treatment at 28 Days
Description: R5-R20 assessed by impulse oscillometry after treatment with solithromycin and placebo.
Time Frame: 28 days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: kiloPascals per liter per second
Arm/Group | Solithromycin | Placebo
Number analyzed (Participants) | 3 | 4
kiloPascals per liter per second | 0.31 (0.06) | 0.21 (0.05)

11. Secondary Outcome: COPD Assessment Test (CAT) Scores
Description: COPD Assessment Test (CAT) scores after treatment with solithromycin and placebo.
  score of 0-40 to indicate the impact of the disease, the higher score better outcome
Time Frame: 28 days
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Solithromycin | Placebo
Number analyzed (Participants) | 3 | 4
score on a scale | 16 (4) | 15 (5)

12. Secondary Outcome: The Number of Adult COPD Patients With Treatment-related Adverse Events, as Assessed by CTCAE v4.0.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Solithromycin | Placebo
Number analyzed (Participants) | 5 | 5
Participants | 5 | 0

13. Other Pre Specified Outcome: Exploratory Outcome: Activity of HDAC2 in Sputum Macrophages From Patients, Before and After Treatment With Solithromycin and Placebo.
Time Frame: 28 days
Population: No data collected for this Outcome due to early termination of the trial
Arm/Group | Solithromycin | Placebo
Number analyzed (Participants) | 0 | 0

14. Other Pre Specified Outcome: Exploratory Outcome: Activity of PI3K in Sputum Macrophages From Patients, Before and After Treatment With Solithromycin and Placebo.
Time Frame: 84 days
Population: No data collected for this Outcome due to early termination of the trial
Arm/Group | Solithromycin | Placebo
Number analyzed (Participants) | 0 | 0

15. Other Pre Specified Outcome: Exploratory Outcome: Activity of NF-κB in Sputum Macrophages From Patients, Before and After Treatment With Solithromycin and Placebo.
Time Frame: 28 days
Population: No data collected for this Outcome due to early termination of the trial
Arm/Group | Solithromycin | Placebo
Number analyzed (Participants) | 0 | 0

16. Other Pre Specified Outcome: Exploratory Outcome: Levels of the Serum Biomarker C-reactive Protein Before and After Treatment With Solithromycin and Placebo.
Time Frame: 28 days
Population: No data collected for this Outcome due to early termination of the trial
Arm/Group | Solithromycin | Placebo
Number analyzed (Participants) | 0 | 0

17. Other Pre Specified Outcome: Exploratory Outcome: Levels of Serum Biomarkers Fibrinogen Before and After Treatment With Solithromycin and Placebo.
Time Frame: 28 days
Population: No data collected for this Outcome due to early termination of the trial
Arm/Group | Solithromycin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 28 days for each treatment period
Arm/Group | Solithromycin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/6 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solithromycin (N=6) | Placebo (N=6)
Elevated liver tests (Hepatobiliary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solithromycin (N=6) | Placebo (N=6)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastro-oesophageal reflux (Gastrointestinal disorders) | 2 (2) | 0 (0)
Derranged LFTs (Hepatobiliary disorders) | 1 (1) | 0 (0)
Puffy eyes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations of the trial such as small numbers of subjects analysed or technical problems leading to unreliable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes